CLINICAL TRIAL: NCT06274268
Title: Effect of Sarcopenia on the Occurrence of Toxicity Related to Anti-cancer Treatments. Prospective Cohort Study
Brief Title: Effect of Sarcopenia on the Occurrence of Toxicity Related to Anti-cancer Treatments
Acronym: SARC-ONCO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Metropole Savoie (Other)
Collaborators: Université Savoie Mont Blanc (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHMS23006
Record Dates: First submitted 2024-02-01; First posted 2024-02-23 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Sarcopenia; Oncology; Physical Inactivity; Toxicity Due to Chemotherapy
MeSH Terms: conditions — Sarcopenia; Neoplasms; Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: Prospective cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventionnal (Experimental): "Hand Grip" Dynamometer Chair rise test measurement of impedance SEFI Nutritional Intake Assessment Questionnaire GPAQ questionnaire SARC-F questionnaire
  Interventions: Diagnostic Test: Sarcopenia diagnostic test

INTERVENTIONS:
Diagnostic Test: Sarcopenia diagnostic test — the study-specific measurements for the assessment of sarcopenia (impedancemetry, grip strength and chair rise test) as well as the distribution of actimeters to patients.

SUMMARY:
The goal of this clinical trial is to learn about the effect of sarcopenic status on the occurrence of treatment-related toxicity during the first course of anti-cancer treatment in several types of cancers.

The main question it aims to answer is :

Is sarcopenia a predictive marker for the occurrence of toxicity in the initial phase of cancer treatment?

The evaluation will focus on the body composition of the participants, assessed by impedancemetry, and on their muscular performance by standardized physical tests.

DETAILED DESCRIPTION:
The present study is single-center within the Centre Hospitalier Metropole Savoie, interventional and prospective, and will be carried out in patients suffering from cancer and having received an indication for systemic oncological treatment, in first line,

The inclusion visit (V1) will take place during the first chemotherapy session and will include study-specific measurements for the assessment of sarcopenia (impedancemetry, grip strength and chair rise test) as well as the distribution of actimeters to patients. The duration of these examinations carried out in addition to clinical practice is estimated at 15 minutes and does not involve any particular risks for patients.

Data collection 1 (R1) will be carried out during the second course of chemotherapy, data collection 2 (R2) will be carried out 6 months from the start of treatment, and data collection 3 (R3) at 12 months from the start of treatment. inclusion, based on standardized extraction of the medical file.

An exploratory study will be offered to patients treated in the context of adjuvant or neoadjuvant breast cancer and treated by the AC/PACLITAXEL protocol which will involve a second optional visit (optional V1.1) during the first injection of PACLITAXEL . An optional data collection (R1.1) will take place during the first cycle to collect actimetry data. And an optional data collection (R1.2) will take place 2 weeks after the theoretical end of PACLITAXEL in order to collect on file the grades of neuropathies and toxicities over the interval.

The visits will be carried out as part of the usual patient care.

Apart from the measurement of impedancemetry, grip strength, the chair rise test and actimetry, no other clinical, paraclinical intervention or biological analysis will be induced by the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old
* Patient with a diagnosis of a histologically proven solid malignant tumor with an indication for systemic treatment during initial treatment.
* CT/PET performed within 45 days before initiation of systemic treatment.
* Patient able to sign informed consent for participation in the study
* Patient affiliated to a social security system

Exclusion Criteria:

* History of cancer in the five years preceding inclusion other than localized skin or cervical cancers.
* Patient with cancer not requiring systemic treatment.
* Pregnant women.
* Patient with a pace maker or defibrillator
* Patient deprived of liberty or benefiting from a legal protection measure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2024-06-24 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Event-free survival according to sarcopenic statut | Day 1 of the first treatment cycle to Day 1 of the second treatment cycle, approx. 4 weeks
  Event-free survival will be defined as the time from the date of the experimental visit to the date of the first documented dose-limiting toxicity. Participants who will not experience an event as of the time of data cut-off (beginning of the second cycle of treatment) or who stopped study participation before the end of the follow-up, will be right-censored. The measure will be analyzed using a COX multivariate model with event incidence rate as dependant variable and the sarcopenia statut as independent variable.

SECONDARY OUTCOMES:
Event-free survival according to the link between: 1/ the dose/lean mass ratio and 2/ body composition and the occurrence of adverse events linked to treatment. | Day 1 of the first treatment cycle to Day 1 of the second treatment cycle, approx. 4 weeks
  Event-free survival will be defined as for the primary outcome. The measure will be analyzed using a COX multivariate model with event incidence rate as dependant variable and the sarcopenia statut, the dose/lean mass ratio and the body composition indices (fat free mass (kg) and fat mass (kg)), as independent variables.
Progression free-survival | 12 months
  Progression : ≥ 20% increase in the sum of the diameters of the target lesions compared to the smallest sum of the diameters observed during the study (NADIR), including the baseline visit. In addition to this relative increase of 20%, this sum must increase by at least 0.5 cm. Note: the appearance of one or more new lesions is also considered progression.
  Progression-free survival will be defined as the time from the date of the experimental visit to the date of the first documented progression.
  Participants who will not experience a progression as of the time of data cut-off (end of 12 month follow-up) or who stopped study participation before the end of the follow-up, will be right-censored. The measure will be analyzed using a COX multivariate model with progression incidence rate as dependant variable and the sarcopenia statut, the dose/lean mass ratio and the body composition indices (fat free mass (kg) and fat mass (kg)), as independent variables.
Overall survival | 12 months
  Overall survival will be defined as the time from the date of the experimental visit to the date of death (irrespective of cause).
  Participants who will be alive at the time of data cut-off (end of 12 month follow-up) or who stopped study participation before the end of the follow-up, will be right-censored. The measure will be analyzed using a COX multivariate model with death incidence rate as dependant variable and the sarcopenia statut, the dose/lean mass ratio and the body composition indices (fat free mass (kg) and fat mass (kg)), as independent variables.
Objective response rate at 6 and 12 months | 6 and 12 months
  For metastatic or locally advanced patients, ORR will be defined as the percentage of subjects with Complete response (CR) or Partial response (PR), according to RECIST v1.1. For patients in adjuvant/neoadjuvant treatment, ORR will be defined as the percentage of subjects with confirmation of no relapse by the investigator based on the analysis of an imaging examination. ORR will be analyze as dependent variable in a logistic regression model including sarcopenia statut, the dose/lean mass ratio and the body composition indices (fat free mass (kg) and fat mass (kg)) as independent variables.
Number of patients classified as sarcopenic by BIA method and CT method. | at baseline
  Taking CT evaluation as the reference method, evaluate: the sensitivity, specificity, negative and positive predictive value of BIA to detect sarcopenia.
Exploratory: Event-free survival during PACLITAXEL protocol | 14 weeks after initiation of paclitaxel protocol
  Event-free survival will be defined as the time from the date of the first PACLITAXEL injection to the date of the first documented dose-limiting toxicity. Participants who will not experience an event as of the time of data cut-off (14 weeks after the initiation of PACLITAXEL protocol) or who stopped study participation before the end of the follow-up, will be right-censored. The measure will be analyzed using a COX multivariate model with event incidence rate as dependent variable and the sarcopenia statut as independent variables.
Exploratory: Level of spontaneous activity measurement by accelerometry (m.s-2). | Day 1 of the first treatment cycle to Day 1 of the second treatment cycle, approx. 4 weeks.
  Compare, according to sarcopenic status and the occurrence of treatment-related adverse events, the level of spontaneous physical activity by accelerometry over the treatment 1/treatment 2 interval.
Exploratory: RCB-based objective response rate at 6 and 12 months | At the time of surgical mastectomy
  For patients with triple negative or HER2 positive breast tumor, ORR will be defined as the percentage of subjects with RCB (residual cancer burden) 0, I or II according to histological analysis of the surgical specimen. ORR will be analyze as dependent variable in a logistic regression model including sarcopenia statut, the dose/lean mass ratio and the body composition indices (fat free mass (kg) and fat mass (kg)) as independent variables.

CONTACTS AND LOCATIONS:
Overall Officials: Aurelie FILLON, Principal Investigator — Centre Hospitalier Metropole Savoie
Locations (1):
- Centre Hospitalier Metropole Savoie, Chambéry, France

IPD SHARING:
Plan to Share IPD: No